CLINICAL TRIAL: NCT06046911
Title: Effects of Tai Chi on Postural Balance and Quality of Life Among Elderly With Gait Disorders in China
Brief Title: Effects of Tai Chi on Postural Balance and Quality of Life in the Elderly With Gait Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, XU FAN, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Xu Fan
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Gait Disorder; Postural Balance
Keywords: Tai Chi; Balance; Gait; Quality of life; Muscle strength
MeSH Terms: conditions — Mobility Limitation | interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: In this experiment, the experimental group will practice Yang Style Tai Chi.The control group will be the daily activity group, maintaining daily activities such as walking. There are males and females in each parallel group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi group (Experimental): The intervention was 12 weeks of Yang-style Tai Chi, three times a week.
  Interventions: Other: Tai Chi
- Daily activity group (Experimental): The daily activity group mainly maintained daily activities, such as walking and stretching, three times a week for 12 weeks.
  Interventions: Other: Daily activity group

INTERVENTIONS:
Other: Tai Chi — In this study, Tai Chi has a total of 24 movements, which are connected step by step according to the principles of sports training.
  Arms: Tai Chi group
Other: Daily activity group — The daily activity group does not receive special intervention, and the subjects must maintain their daily habits and complete the 12-week test.
  Arms: Daily activity group

SUMMARY:
The goal of this intervention study was to test balance ability and quality of life in older adults with gait problems. The main questions it aims to answer are: 1. Can the balance ability of elderly people with gait disorders be improved through Tai Chi intervention? 2. Whether Tai Chi intervention can improve the quality of life of elderly people with gait disorders.

Participants will be divided into an experimental group and a control group. The experimental group will undergo 12 weeks of Tai Chi intervention, while the control group will maintain daily habits, including simple walking or stretching activities.

DETAILED DESCRIPTION:
The inclusion criteria for potential participants were as follows:

Age ≥ 60 years old Have mild gait problems Can walk independently No Tai Chi training experience or exercise habits

The exclusion criteria for potential participants were as follows:

Age <60 years old No obvious problems with gait walking with tools Have experience in Tai Chi intervention within three months hearing loss

Outcomes measured: balance, gait, muscle strength, mobility, fall rate, quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years old Have mild gait problems Can walk independently No Tai Chi training experience or exercise habits

Exclusion Criteria:

* Age <60 years old No obvious problems with gait walking with tools Have experience in Tai Chi intervention within three months hearing loss

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Effects of 12 weeks of Tai Chi intervention on balance ability in the elderly | The balance ability of the elderly was tested before the intervention, after 6 weeks of intervention, and at 12 weeks
  The main test method is the single-leg eyes-closed test
Effects of 12 weeks of Tai Chi intervention on gait speed of the elderly | The gait speed of the elderly was tested before the intervention, after 6 weeks of intervention, and at 12 weeks
  Gait speed measurement mainly uses the four-meter walking test
Effects of 12 weeks of Tai Chi intervention on gait skills | The gait skills of the elderly were tested before the intervention and at 6 and 12 weeks after the intervention
  Gait skill measurement mainly uses the figure-8 walking test
Effects of 12-week Tai Chi intervention on mobility of the elderly | The Mobility of the elderly was tested before the intervention, after 6 weeks of intervention, and at 12 weeks
  Time Up and Go measures mobility
Effects of 12 weeks of Tai Chi intervention on upper limb muscle strength in the elderly | The upper limb muscle strength of the elderly was tested before the intervention, after 6 weeks of intervention, and at 12 weeks
  Grip strength test upper limb muscle strength
Effects of 12 weeks of Tai Chi intervention on lower limb muscle strength in the elderly | The lower limb muscle strength of the elderly was tested before the intervention, after 6 weeks of intervention, and at 12 weeks
  30s chair test to measure lower limb muscle strength
Effect of 12-week Tai Chi intervention on fall risk in the elderly | The Fall risk of the elderly was tested before the intervention, after 6 weeks of intervention, and at 12 weeks
  Time Up and Go measures Fall risk
Effects of 12-week Tai Chi intervention on the quality of life of the elderly | The Quality of life of the elderly was tested before the intervention, after 6 weeks of intervention, and at 12 weeks
  Measured using Questionnaire, 36-Item Short Form Surve (SF-36) Scale

CONTACTS AND LOCATIONS:
Overall Officials: Fan Xu, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Binhe Sports Center, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borowicz A, Zasadzka E, Gaczkowska A, Gawlowska O, Pawlaczyk M. Assessing gait and balance impairment in elderly residents of nursing homes. J Phys Ther Sci. 2016 Sep;28(9):2486-2490. doi: 10.1589/jpts.28.2486. Epub 2016 Sep 29. PMID 27799676
- [Background] Chang JH, Koo M, Wu SW, Chen CY. Effects of a 12-week program of Tai Chi exercise on the kidney disease quality of life and physical functioning of patients with end-stage renal disease on hemodialysis. Complement Ther Med. 2017 Feb;30:79-83. doi: 10.1016/j.ctim.2016.12.002. Epub 2016 Dec 7. PMID 28137531
- [Background] Taylor-Piliae RE, Haskell WL, Waters CM, Froelicher ES. Change in perceived psychosocial status following a 12-week Tai Chi exercise programme. J Adv Nurs. 2006 May;54(3):313-29. doi: 10.1111/j.1365-2648.2006.03809.x. PMID 16629916
- [Background] Huang SL, Hsieh CL, Wu RM, Tai CH, Lin CH, Lu WS. Minimal detectable change of the timed "up & go" test and the dynamic gait index in people with Parkinson disease. Phys Ther. 2011 Jan;91(1):114-21. doi: 10.2522/ptj.20090126. Epub 2010 Oct 14. PMID 20947672
- [Background] Ke XH, Huang DB, Li YY, Li XM, Guo JH, Guo MM, Yu SX, Ma SC, Jiang C, Lin ZH. Effects of 12 weeks of Tai Chi Chuan intervention on the postural stability and self-reported instability in subjects with functional ankle instability: Study protocol for a randomized controlled trial. Front Neurol. 2022 Sep 21;13:923669. doi: 10.3389/fneur.2022.923669. eCollection 2022. PMID 36212637
- [Background] Perez-Cruzado D, Gonzalez-Sanchez M, Cuesta-Vargas AI. Parameterization and reliability of single-leg balance test assessed with inertial sensors in stroke survivors: a cross-sectional study. Biomed Eng Online. 2014 Aug 30;13:127. doi: 10.1186/1475-925X-13-127. PMID 25174611
- [Background] Soke F, Demirkaya S, Gulsen C, Yavuz N, Karakoc S, Ozcan Gulsen E, Yilmaz O, Kocer B, Kurtulus Aydin F, Yucesan C. The figure-of-eight walk test is a reliable and valid test for assessing walking skill in people with multiple sclerosis. Mult Scler Relat Disord. 2022 Nov;67:104099. doi: 10.1016/j.msard.2022.104099. Epub 2022 Aug 9. PMID 35969935
- [Background] Taylor-Piliae RE, Hoke TM, Hepworth JT, Latt LD, Najafi B, Coull BM. Effect of Tai Chi on physical function, fall rates and quality of life among older stroke survivors. Arch Phys Med Rehabil. 2014 May;95(5):816-24. doi: 10.1016/j.apmr.2014.01.001. Epub 2014 Jan 17. PMID 24440643
- See also: Assessment of the 4-meter walk test test-retest reliability and concurrent validity and its correlation with the five sit-to-stand test in chronic ambulatory stroke survivors — https://doi.org/10.1016/j.gaitpost.2023.01.014